CLINICAL TRIAL: NCT05259085
Title: A Phase 1, Open-Label, Multiple-Dose, Parallel Study to Determine the Effect of Hepatic Impairment on the Pharmacokinetics, Safety, and Tolerability of ALXN2050 in Adult Participants
Brief Title: Study of ALXN2050 in Participants With Hepatic Impairment
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision.
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ALXN2050-HV-109
Record Dates: First submitted 2020-11-05; First posted 2022-02-28 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-02

CONDITIONS: Impaired Hepatic Function; Healthy
Keywords: Pharmacokinetics; Safety; Factor D inhibitor; ALXN2050
MeSH Terms: interventions — rhoA GTP-Binding Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ALXN2050 (Experimental): Cohort 1: Mild IHR Cohort 2: Moderate IHR Cohort 3: Severe IHR Cohort 4: Healthy Control
  Participants will receive ALXN2050
  Interventions: Drug: ALXN2050

INTERVENTIONS:
Drug: ALXN2050 — ALXN2050 (120 milligrams) will be administered orally twice daily on Days 1 through 3, with an additional dose (120 milligrams) administered orally on the morning of Day 4.
  Other Names: ACH-0145228 (formerly)

SUMMARY:
This study will investigate the impact of impaired hepatic function (IHF) on the plasma pharmacokinetics of ALXN2050 in order to provide dosing recommendations for future indications in individuals with varying degrees of IHF.

DETAILED DESCRIPTION:
The study will initiate (Part 1) with participants with mild IHF (Cohort 1) and moderate IHF (Cohort 2) and their matched healthy control participants (Cohort 4). Cohort 1 will be enrolled first, and following an adequate safety review, enrollment for Cohort 2 will begin. Following data review, the study may proceed (Part 2) with participants with severe IHF (Cohort 3) if deemed necessary.

ELIGIBILITY:
Inclusion Criteria:

1. Body weight must be at least 50.0 kilograms (kg) and body mass index (BMI) within the range of 18.0 - 40.0 kg/meter squared (inclusive) at the time of signing the informed consent.
2. Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
3. Must agree to receive prophylactic antibiotics to mitigate the potential risk of meningococcal infection.

   Participants with Impaired Hepatic Function
4. Aside from IHF, sufficiently healthy for study participation based upon medical history, physical examination, neurological examination, laboratory tests, vital signs, and electrocardiograms (ECGs).
5. Score on the Child-Pugh scale at screening as follows:

   * Mild: Class A (Child-Pugh score ≥5 and ≤6); or
   * Moderate: Class B (Child-Pugh score ≥7 and ≤9); or
   * Severe: Class C (Child-Pugh score ≥10 and ≤15).
6. Diagnosis of chronic (>6 months), stable (no acute episodes of illness within the previous 1 month due to deterioration in hepatic function) hepatic insufficiency.
7. Must be on a stable medication regimen. Concomitant medications must be approved by Alexion unless presented in the list of common concurrent medications for participants with IHF.
8. Cirrhosis, as evidenced by parenchymal liver disease by biopsy (histological diagnosis), imaging test, or other suitable imaging study, due to chronic hepatitis C virus (HCV) infection, chronic hepatitis B infection, cryptogenic, alcohol abuse, or non-alcoholic steatohepatitis.
9. No evidence of hepatocellular carcinoma as documented by imaging within 6 months prior to the first dose of study intervention.

   Matched Healthy Control Participants with Normal Hepatic Function
10. Must match the sex (similar ratio) and race (similar ratio of white and non-white) of participants with IHF; age must be within ± 10 years and BMI must be within ± 20% of participants with IHF at screening.
11. Healthy as determined by medical evaluation including medical history, physical examination, neurological examination, laboratory tests, vital signs, and ECGs.

Exclusion Criteria:

1. History or presence of seizures, head injury, head trauma, or any other brain disorder.
2. History of procedures that could alter absorption or excretion of orally administered drugs.
3. History of meningococcal infection or a first-degree relative with a history of meningococcal infection.
4. Body temperature ≥38.0°Celcius at screening or check-in or history of febrile illness or other evidence of infection, systemic or otherwise, within 14 days prior to the first dose of study intervention.
5. Classical pathway hemolysis results outside the reference ranges at screening, unless approved by Alexion.
6. Significant blood loss or donation of blood within 3 months prior to the first dose of study intervention, donation of plasma within 30 days prior to the first dose of study intervention, receipt of blood products within 6 months prior to first dose of study intervention, or receipt of a vaccine within 30 days prior to the first dose of study intervention.
7. Current enrollment or past participation within the last 30 days (or 5 half-lives, whichever is longer) prior to the first dose of study intervention in the current clinical study or any other clinical study involving an investigational study intervention or any other type of medical research.
8. Pregnant or lactating.
9. History or presence of drug or alcohol abuse within 6 months prior to the first dose of study intervention, current tobacco user, or positive results for alcohol and/or drug screen at screening or check-in.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-04-07 (Actual); Primary Completion 2024-08-12 (Actual); Study Completion 2024-08-12 (Actual)

PRIMARY OUTCOMES:
Area Under The Concentration-time Curve From Time 0 To The 12-hour Time Point (AUC0-12) Of Plasma ALXN2050 After Steady-state | Up to 72 hours postdose
Maximum (Peak) Steady-state Plasma Concentration Of ALXN2050 (Cmax,ss) | Up to 72 hours postdose
Time To Reach Maximum (Peak) Plasma Concentration Following ALXN2050 Administration At Steady-state (Tmax,ss) | Up to 72 hours postdose

SECONDARY OUTCOMES:
Number Of Participants Receiving ALXN2050 With Treatment-emergent Adverse Events | Day 1 (postdose) through follow-up (30 [+/- 2] days after last study drug administration)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Research Site, Hialeah, Florida
  - Research Site, Orlando, Florida

IPD SHARING:
Plan to Share IPD: No